CLINICAL TRIAL: NCT04953624
Title: Detection of Appetite and Analysis of Related Factors in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Appetite and Related Factors in Patients With ALS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020399
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CNAQ≤28: ALS patients with CNAQ ≤ 28
  Interventions: Diagnostic Test: Appetite rating scale CNAQ
- CNAQ>28: ALS patients with CNAQ > 28
  Interventions: Diagnostic Test: Appetite rating scale CNAQ

INTERVENTIONS:
Diagnostic Test: Appetite rating scale CNAQ — Chinese version of Appetite rating scale CNAQ

SUMMARY:
Chinese cnaq scale was used to evaluate the appetite changes of Chinese ALS patients; Objective to investigate the related factors of appetite changes in ALS patients; Objective to investigate the effect of anorexia on the progression and survival of ALS patients.

DETAILED DESCRIPTION:
1. With the consent of the original author, the scale was translated and back translated, and the Chinese version of the scale was determined after communication and confirmation with the original author.
2. Cnaq was used to measure the appetite of the patients, and hads was used to measure the anxiety and depression of the patients;
3. Analyze the proportion of loss of appetite in ALS group, compare the differences of clinical characteristics such as ALSFRS-R score, weight, BMI value, cognitive status such as ECAs score between patients with loss of appetite and patients without loss of appetite in ALS group, and conduct correlation analysis.
4. The patients were followed up every three months until they were unable to eat or end-point events (invasive ventilator or death), and the correlation between cnaq and disease progression and survival was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients diagnosed as probable, or definite according to the revised El Escorial criteria

Exclusion Criteria:

* there are other chronic consumption diseases such as severe digestive system diseases, thyroid diseases, diabetes and so on.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ALS patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R score | 3 months
ALSFRS-R score | 6 months
ALSFRS-R score | 12 months
Food intake | 3 months
  Inability to eat
Food intake | 6 months
  Inability to eat
Food intake | 12 months
  Inability to eat
invasive ventilator or death | 3 months
  end point events
invasive ventilator or death | 6 months
  end point events
invasive ventilator or death | 12 months
  end point events

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes